CLINICAL TRIAL: NCT04505748
Title: Is Serum Gentamicin Concentration Modified With Autologous Cell-saved Blood Transfusion After Total Knee Arthroplasty Using Tranexamic Acid: A Randomized Control Trial
Brief Title: Is Self-transfusion Safe After Total Knee Arthroplasty in Terms of Nephrotoxicity of Gentamicin From Bone Cement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Alexandroupolis (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Panagiotis Touzopoulos, Consultant of Orthopaedic Surgery, University Hospital, Alexandroupolis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 80/27-01-2017
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Arthroplasty Complications; Total Knee Arthroplasty
Keywords: gentamicin; self-transfusion; blood loss; toxicity; total knee arthoplasty
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-transfusion group (Experimental): Patients to whom a self-transfusion device has been used after total knee arthroplasty.
  Interventions: Device: Self-transfusion device
- Control group (No Intervention): Patients to whom conventional drains have been used after total knee arthroplasty.

INTERVENTIONS:
Device: Self-transfusion device — The Transfusion filter set for salvaged blood (Summit Medical Ltd, Gloucestershire, UK) has been randomly used in 20 patients postoperatively. Patients, who received autologous blood, transfused with the collected amount of blood, only once, 6h postoperatively
  Arms: Self-transfusion group

SUMMARY:
Considering that the high local concentration of antibiotic from bone cement is delivered intravenously through the self-transfusion process, systematic toxicity has never been evaluated. In addition, the effectiveness of self-transfusion with the routine concomitant use of other modern blood-salvage strategies, like tranexamic acid, should be also assessed. Therefore we performed a randomized study to assess: 1) the safety of self-transfusion in TKA by comparing the gentamicin concentrations resulting from the use or not of autologous blood transfusion. 2) the efficacy of self-transfusion in TKA, with the concomitant administration of tranexamic acid.

The serum concentration of aminoglycosides has been measured in two groups of 20 patients each, after TKA, according to the use of self-transfusion. Hemoglobin, renal function and calculated blood loss were compared at several time points between groups.

ELIGIBILITY:
Inclusion Criteria:

* end-stage of knee osteoarthritis, who scheduled for unilateral primary TKA in our department

Exclusion Criteria:

* patients who had been treated with gentamicin within the past 10 days
* known allergies against the bone cement
* estimated glomerular filtration rate (eGFR) <30ml/minute
* previous nephrectomy and history of renal transplant
* contraindications against tranexamic acid

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Gentamicin serum concentration | Postoperatively at: 1 hour, 6 hours, 7 hours, 24 hours and 48 hours.
  using a quantitative fluorescent polarizing immunoassay (FPIA) in the Biochemical analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Verceridis, PhD, Study Director — Associate Professor of Orthopedics, School of Medicine, Democritus University of Thrace, Greece
Locations (1):
- University General Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrick BN, Rivey MP, Allington DR. Acute renal failure associated with vancomycin- and tobramycin-laden cement in total hip arthroplasty. Ann Pharmacother. 2006 Nov;40(11):2037-42. doi: 10.1345/aph.1H173. Epub 2006 Oct 10. PMID 17032907
- [Background] Parvizi J, Saleh KJ, Ragland PS, Pour AE, Mont MA. Efficacy of antibiotic-impregnated cement in total hip replacement. Acta Orthop. 2008 Jun;79(3):335-41. doi: 10.1080/17453670710015229. PMID 18622836
- [Result] de Klaver PA, Hendriks JG, van Onzenoort HA, Schreurs BW, Touw DJ, Derijks LJ. Gentamicin serum concentrations in patients with gentamicin-PMMA beads for infected hip joints: a prospective observational cohort study. Ther Drug Monit. 2012 Feb;34(1):67-71. doi: 10.1097/FTD.0b013e31823d7b89. PMID 22249345
- [Derived] Touzopoulos P, Arvanitidis K, Filidou E, Tilkeridis K, Karanikas M, Kolios G, Ververidis A. Is serum gentamicin concentration modified with autologous cell-saved blood transfusion after total knee arthroplasty using tranexamic acid? A randomised control trial. Orthop Traumatol Surg Res. 2021 May;107(3):102794. doi: 10.1016/j.otsr.2020.102794. Epub 2020 Dec 14. PMID 33333277